CLINICAL TRIAL: NCT00597415
Title: A Double-Blind, Placebo-Controlled, Randomized, Crossover Pilot Study of the Efficacy of Celecoxib 200 mg QD in Relieving Pain and Walking Dysfunction in Osteoarthritis of the Knee.
Brief Title: Efficacy of Celecoxib 200mg in Relieving Pain and Walking Dysfunction in Osteoarthritis of the Knee
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Nora G. Singer MD, University Hospitals Case Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Pfizer walking model; UH IRB 06-04-41
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2008-01-18 (Estimated); Status verified 2007-12

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; Knee pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A 1 (Placebo Comparator): A 1=placebo
  Interventions: Drug: placebo
- A 2 (Active Comparator): A 2=celecoxib
  Interventions: Drug: celecoxib

INTERVENTIONS:
Drug: celecoxib — celecoxib 200mg
  Other Names: Celebrex
  Arms: A 2
Drug: placebo — placebo
  Other Names: inactive capsule
  Arms: A 1

SUMMARY:
The purpose of this study is to compare the efficacy of celecoxib versus placebo in delaying the onset of pain and improving walking function in subjects with knee Osteoarthritis

DETAILED DESCRIPTION:
We have developed a walking model that safely and reproducibly induces pain in subjects with knee OA in a manner that permits the comparison of the effect of different therapies on pain control. In a previous study, we demonstrated that a self-paced 20 minute walk followed by a one-hour rest and a second coordinator-paced 20-minute walk was well tolerated and generated moderate to severe pain in all participants within the time frame of the walk. We will now use this model, but with a crossover design to test the efficacy of celecoxib compared to placebo for the control of knee pain and improvement of walking function.

ELIGIBILITY:
Inclusion Criteria:

* If female and of childbearing potential, must be using adequate contraception since last menses and will use adequate contraception during the study,
* Diagnosed as having OA of the knee
* Functional Capacity Classification of I-II (FCC)
* If on active analgesic or anti-inflammatory pain medication, must have VAS pain score>=30mm in signal knee related to walking on a flat surface within the previous 48 hours. Subjects who are not taking any pain medication must have a VAS pain score>=40mm in the signal knee
* At baseline visit, must have a history of pain in the signal knee>=40mm when walking on the flat within the previous 48 hours.
* In the Investigator's opinion, the patient requires and is eligible for therapy with an anti-inflammatory analgesic.
* If on an NSAID or analgesic, patient must have completed a washout period prior to baseline assessments that is a minium of five half lives.
* The patient has provided written informed consent before undergoing any study procedures.

Exclusion Criteria:

* Diagnosed as having inflammatory arthritis or acute trauma at the index joint.
* Another painful condition that would interfere with his/her ability to walk or to make reasonable assessments of their pain.
* Received an injection of corticosteroid into the signal knee within 3 months; or with a hyaluronan produce in the signal knee within the previous 6 months.
* Requires the use of a cane or other assistive device to complete the walk.
* Known cardiovascular disease which has been symptomatic in the past 12 months
* History of blood clots or is at any increased risk for blood clotting.
* Asthma or any breathing condition which would preclude walking briskly for 20 consecutive minutes or 40 minutes total.
* Has taken any NSAIDs, COX-2 inhibitors, or any analgesic, with the exception of the rescue acetaminophen, within two days prior to Visit 2
* Active malignancies or any type or a malignancy that has recurred within 5 years before enrollment.
* Diagnosed as having or has been treated for esophageal, gastric, pyloric channel, duodenal ulceration within 90 days
* Active GI disease, a chronic or acute renal or hepatic disorder, or a significant coagulation defect.
* Any chronic illness or laboratory abnormalities considered to be clinically significant.
* Received any investigational medication within 30 days
* Known hypersensitivity to celecoxib, NSAIDs, to sulfonamides
* Use of the following drugs:

  1. NSAIDs or COX-2 specific inhibitors
  2. Analgesics except rescue medication within 24 hours of a study visit
  3. Anticoagulants
  4. Lithium
  5. Glucosamine or chondroitin sulfate are excluded unless on stable dose for at least 3 months

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-12; Primary Completion 2008-02 (Estimated); Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the time to onset of moderate and severe pain. The mean change in time to onset of moderate and sever pain between the first and second walks will be compared using paired t-tests. | Visits 2 and 3

SECONDARY OUTCOMES:
Secondary endpoints are the distance to onset of moderate to sever pain the the percent responders in each group. Thirty subjects will be studied in this randomized, placebo-controlled, double-blind crossover study. | Visits 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Nora G Singer, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Beachwood, Ohio, United States